CLINICAL TRIAL: NCT03289897
Title: Non-invasive Rapid Assessment of Non-alcoholic Fatty Liver Disease (NAFLD) Using Magnetic Resonance Imaging With LiverMultiScan (RADIcAL1)
Brief Title: Non-invasive Rapid Assessment of NAFLD Using Magnetic Resonance Imaging With LiverMultiScan
Acronym: RADIcAL1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perspectum (Industry)
Collaborators: University of Coimbra (Other); University Hospital Ulm (Other); Leiden University Medical Center (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); University Hospital Southampton NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); NHS Greater Glasgow and Clyde (Other); Glasgow Royal Infirmary (Other); Ninewells Hospital (Other); Royal Infirmary of Edinburgh (Other); St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PJM124
Record Dates: First submitted 2017-09-05; First posted 2017-09-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; NAFLD; Metabolic Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm-LiverMultiScan (Experimental): Patients will be scanned using the LiverMultiScan. Follow-up will be determined by the results of the scan.
  Interventions: Diagnostic Test: LiverMultiScan
- Control Arm (No Intervention): Standard of care as per guidelines of the local centre

INTERVENTIONS:
Diagnostic Test: LiverMultiScan — LiverMultiScan is an imaging technique which is able to identify early liver disease.
  Arms: Study Arm-LiverMultiScan

SUMMARY:
A multi-centre randomised controlled trial to determine the implementation and health care cost of LiverMultiScan vs. routine methodical assessment (standard care) of Non-alcoholic fatty liver disease (NAFLD) across several European countries.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a condition associated with obesity, insulin resistance and heart disease. Research has shown that fatty liver (steatosis) can lead to a spectrum of diseases including low grade inflammation (steatohepatitis or non-alcoholic steatohepatitis (NASH)), cirrhosis or liver failure.

The current method used to diagnose liver dysfunction and failure is with percutaneous liver biopsy. This is painful and is not without risk, as the liver is a highly vascular organ. Even with ultrasound guidance, it carries a 1:1000 risk of serious adverse events (e.g. bleeding, infection, bowel perforation). As a result of these factors, liver biopsy is not used in all patients with suspected NAFLD/ NASH unless moderate to severe liver disease is presented or other liver disease need to be excluded. Various diagnostic pathways have arisen, but in the absence of a clearly non-invasive discriminatory test that can stratify normal liver, simple steatosis, steatohepatitis and cirrhosis, there is no standardised pathway.

LiverMultiScan has been tested against liver biopsy and has been shown to be the first imaging test that can identify early liver disease and predict clinical outcomes accurately. LiverMultiScan has recently been CE-Marked and FDA-cleared, so is available for clinical use, but as a new test, it is not yet widely established in clinical practice. This study will utilise LiverMultiScan and see if it can be the basis of a viable diagnostic pathway in EU healthcare systems by adopting it in different EU countries, and determining the economic costs and benefits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-75 years, due to undergo evaluation for suspected non-alcoholic fatty liver disease
* Presence of:

  * elevated liver function tests (ALT, AST or GGT ≥ 1.5 x upper limit of normal and ≤ 5 x upper limit of normal)

OR

* imaging suggestive of Fatty liver disease.

OR

Presence of ≥ 3 of the following criteria:

1. insulin resistance or type 2 diabetes mellitus
2. obesity (BMI > 30 or waist-to-hip ratio > 1.00 for men / > 0.85 for women)
3. hypertension (≥ 130/85 mmHg)
4. elevated triglycerides (≥ 1.7 mmol/l)
5. low HDL-cholesterol (< 1.05 mmol/l for men / < 1.25 mmol/l for women)

   * Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (inc pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Patients with proven liver disease other than NAFLD.
* Liver transplantation
* Patients that present with clinical signs of chronic liver failure (variceal bleeding, ascites, overt encephalopathy)
* Pregnancy
* Alcohol over-use/ abuse as determined by local guidelines
* Patient with known malignant liver tumours and those with any malignancy with life expectancy < 36 months
* Heart failure NYHA stages II-IV
* Severe mental illness
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
To investigate whether the introduction of LiverMultiScan as a standardised diagnostic test for liver disease can prove a cost-effective method in different EU territories. | 1 year
  Proportion of patients with suspected NAFLD incurring liver related hospital consultations and/or liver biopsies, from the date of randomisation to the end of the study follow-up.

SECONDARY OUTCOMES:
Patient satisfaction: questionnaire | 1 year
  Patient feedback from patient satisfaction questionnaire, at baseline, and all follow-up visits to the end of the study.
Certainty of diagnosis | 1 year
  Certainty of diagnosis is defined as binary (yes/no vs. unlikely/probable) at baseline and all follow-up visits to the end of the study.
Frequency of diagnosis | 1 year
  Frequency of diagnosis is defined as binary (yes/probable vs. no/unlikely) at baseline and all follow-up visits to the end of the study.
Time to diagnosis | 1 year
  Time from randomisation to diagnosis by the physician, as recorded at final follow-up visit.
Measure resource use | 1 year
  Rates of liver related outpatient investigations/consultations/hospital admissions per 400 patients during the study.
Cost effectiveness of LiverMultiScan | 1 year
  Cost of LiverMultiScan based on randomised comparison.
Personnel skills required for diagnosis | 1 year
  Percentage of total consultations performed by a specialist, at each specialist medical category, from date of randomisation to end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Dollinger, MD, Principal Investigator — University Hospital Ulm; Dimitar Tonev, MD, Principal Investigator — Perspectum Diagnostics
Locations (11):
- University Hospital Ulm, Ulm, Baden-Wurttemberg, Germany
- Leiden University Medical Center, Leiden, South Holland, Netherlands
- University of Coimbra, Coimbra, Centro, Portugal
- United Kingdom (8):
  - Southampton University Hospital, Southampton, Hampshire
  - Aintree Hospital, Liverpool, Merseyside
  - Ninewells Hospital, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - King's College Hospital, London
  - St George's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- [Derived] Tonev D, Shumbayawonda E, Tetlow LA, Herdman L, French M, Rymell S, Thomaides-Brears H, Caseiro-Alves F, Castelo-Branco M, Ferreira C, Coenraad M, Lamb H, Beer M, Kelly M, Banerjee R, Dollinger M; RADIcAL1. The Effect of Multi-Parametric Magnetic Resonance Imaging in Standard of Care for Nonalcoholic Fatty Liver Disease: Protocol for a Randomized Control Trial. JMIR Res Protoc. 2020 Oct 26;9(10):e19189. doi: 10.2196/19189. PMID 33104014